CLINICAL TRIAL: NCT00366080
Title: An Open Label, Dose Escalation Study With A Double Blind Randomised Placebo Controlled Withdrawal To Examine The Effects Of The Histamine H3 Antagonist GSK189254 In Patients With Narcolepsy.
Brief Title: Effectiveness Of The Drug GSK189254 In Treating Patients With Narcolepsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated based on the interim results of a futility test.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H3A106104
Record Dates: First submitted 2006-08-17; First posted 2006-08-18 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Narcolepsy
Keywords: GSK189254 H3 Histamine Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — 6-((3-cyclobutyl-2,3,4,5-tetrahydro-1H-3-benzazepin-7-yl)oxy)-N-methyl-3-pyridinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK189254

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of the drug GSK189254 in treating patients with narcolepsy.

ELIGIBILITY:
Inclusion criteria:

* Narcolepsy patients
* Body mass index between 18 - 32 kg/m2
* Females may be of child bearing or non-child bearing potential.
* Agreement to refrain from driving or operating heavy machinery for the duration of the study.
* Must be able to withdraw from medication for the treatment of daytime sleepiness and must not be living on their own.

Exclusion criteria:

* History or presence of major psychiatric disorder or depression.
* History of significant head trauma in the previous 12 months.
* Participation in a clinical trial in the previous 3 months.
* Patient has significant and recent (within 1 year) history of drug or alcohol abuse.
* Patient is pregnant or breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Sleep latency (in minutes), as measured by the Maintenance of Wakefulness Test (MWT), at the end of the DBP | Day 42
  Sleep latency was measured at the end of DBP (Day 42) by an extended version of the MWT which was used to measure the ability of a participant to remain awake. The MWT consisted of four 40-minutes trails performed at two hour intervals and the main MWT score was mean sleep latency (arithmetic mean of the four 40-minutes trials). Trials were ended after 40 minutes if no sleep occurred, or after unequivocal sleep, defined as three consecutive epochs of stage 1 sleep, or one epoch of any other stage of sleep. Least square mean was used to present the value for adjusted mean.

SECONDARY OUTCOMES:
Change from baseline in Sleep latency (minutes), as measured by the MWT for the OLP | Baseline (Day -1) and Day 28
  Sleep latency was measured for OLP (Day 28) by an extended version of the MWT which was used to measure the ability of a participant to remain awake. The MWT consisted of four 40-minutes trails performed at two hour intervals and the main MWT score was mean sleep latency (arithmetic mean of the four 40-minutes trials). Trials were ended after 40 minutes if no sleep occurred, or after unequivocal sleep, defined as three consecutive epochs of stage 1 sleep, or one epoch of any other stage of sleep. Baseline was defined at Visit 1 (Day -1). Change from baseline was calculated by subtracting the value on Day -1 minus the value on Day 28.
Change from End of OLP (Day 28) in Sleep latency (minutes), as measured by the MWT to the end of the DBP (Day 42) | Day 28 and Day 42
  Sleep latency was measured by an extended version of the MWT which was used to measure the ability of a participant to remain awake. The MWT consisted of four 40-minutes trails performed at two hour intervals and the main MWT score was mean sleep latency (arithmetic mean of the four 40-minutes trials). Trials were ended after 40 minutes if no sleep occurred, or after unequivocal sleep, defined as three consecutive epochs of stage 1 sleep, or one epoch of any other stage of sleep. Last assessed value of OLP (Day 28) value was used as baseline value for DBP. Change from end of OLP was calculated by subtracting the value on Day 28 minus the value on Day 42. Least square mean was used to present the value for adjusted mean.
Change from Baseline in Frequency of Cataplexy Attacks during the OLP | Baseline (Day -1) up to Day 28
  Narcolepsy was classically described as excessive daytime sleepiness in association with emotionally triggered episodes of muscle weakness, known as cataplexy. Forms of narcolepsy exist without cataplexy which varies in severity from barely perceptible loss of tone of the facial muscles to total collapse. The number of daily cataplexy attacks (frequency) was estimated and recorded in the diary card. Baseline was defined at Visit 1 (Day -1). Change from baseline was calculated by subtracting the value on Day -1 minus the value on Day 1-6, 7-13, 14-20, 21-29.
Change from Baseline in severity of Cataplexy Attacks during the OLP | Baseline (Day -1) up to Day 28
  Narcolepsy was classically described as excessive daytime sleepiness in association with emotionally triggered episodes of muscle weakness, known as cataplexy. Forms of narcolepsy exist without cataplexy which varies in severity from barely perceptible loss of tone of the facial muscles to total collapse. The overall severity of the attacks was rated at the end of each day using a visual analogue scale (VAS) with the following the anchor points: When considering the narcolepsy symptoms for today, overall how severe were the cataplexy Attacks- Not troublesome, e.g. infrequent and/ or had minimal effect on mobility or Very severe, e.g. of high frequency and /or severely debilitating in mobility. Baseline was defined at Visit 1 (Day -1). Change from baseline was calculated by subtracting the value on Day -1 minus the value on Day 1-6, 7-13, 14-20, 21-29.
Change from End of OLP (Day 28) in Frequency of Cataplexy Attacks during the DBP | Day 28 up to Day 42
  Narcolepsy was classically described as excessive daytime sleepiness in association with emotionally triggered episodes of muscle weakness, known as cataplexy. Forms of narcolepsy exist without cataplexy which varies in severity from barely perceptible loss of tone of the facial muscles to total collapse. The number of daily cataplexy attacks was estimated and recorded in the diary card. Last assessed value of OLP (Day 28) value was used as baseline value for DBP. Change from end of OLP was calculated by subtracting the value on Day 28 minus the value on Day 30-35 and 36-42. Least square mean was used to present the value for adjusted mean.
Change from End of OLP (Day 28) in severity of Cataplexy Attacks during the DBP | Day 28 up to Day 42
  Narcolepsy was classically described as excessive daytime sleepiness in association with emotionally triggered episodes of muscle weakness, known as cataplexy. Forms of narcolepsy exist without cataplexy which varies in severity from barely perceptible loss of tone of the facial muscles to total collapse . The number of daily cataplexy attacks was estimated and recorded in the diary card. Last assessed value of OLP (Day 28) value was used as baseline value for DBP. Change from end of OLP was calculated by subtracting the value on Day 28 minus the value on Day 30-35 and Day 36-42. Least square mean was used to present the value for adjusted mean.
Change from Baseline in Severity of Nocturnal Symptoms during the OLP | Baseline (Day -1) up to Day 28
  Participants kept a daily diary card to record the severity of nocturnal narcolepsy symptoms. The overall severity of the nocturnal symptoms was rated at the end of each day using a VAS. In the morning, upon waking and at the time they took their morning dose participants were asked to record the severity of any night time disease symptoms such as hypnagogic hallucinations / sleep paralysis or night terrors using the following question: When considering the sleep you had last night, how troublesome were any dreams, hallucinations or other narcolepsy symptoms such as sleep paralysis- Not troublesome, e.g. hard to remember / not vivid or Very unpleasant, e.g. very vivid and/or of a frightening or disturbing nature. Baseline was defined at Visit 1 (Day -1). Change from baseline was calculated by subtracting the value on Day -1 minus the value on Day 1-6, 7-13, 14-20, 21-29.
Change from End of OLP (Day 28) in Severity of Nocturnal Symptoms during the DBP | Day 28 up to Week 42
  Participants kept a daily diary card to record the severity of nocturnal narcolepsy symptoms. The overall severity of the nocturnal symptoms was rated at the end of each day using a VAS. In the morning, upon waking and at the time they took their morning dose participants were asked to record the severity of any night time disease symptoms such as hypnagogic hallucinations / sleep paralysis or night terrors using the following question: When considering the sleep you had last night, how troublesome were any dreams, hallucinations or other narcolepsy symptoms such as sleep paralysis- Not troublesome, e.g. hard to remember / not vivid or Very unpleasant, e.g. very vivid and/or of a frightening or disturbing nature. Last assessed value of OLP (Day 28) value was used as baseline value for DBP. Change from end of OLP was calculated by subtracting the value on Day 28 minus the value on Day 30-35 and Day 36-42. Least square mean was used to present the value for adjusted mean.
Change from End of OLP (Day 28) on the Epworth Sleepiness Scale (ESS) to the End of DBP (Day 42) | Day 28 up to Day 42
  Subjective sleepiness was measured using ESS, a patient rated measure of excessive daytime sleepiness. ESS was completed by participants at the end of OLP (Day 28) and at the end of DBP (Day 42). Participants estimated their likelihood of falling asleep during 8 normal daily situations (1.Sitting and reading, 2.Watching television, 3.Sitting inactive in public place, such as theatre or meeting, 4.As a passenger in car for an hour without a break, 5.Lying down to rest in the afternoon, 6.Sitting and talking to someone, 7.Sitting quietly after lunch (without alcohol), 8.In a car, while stopped in traffic) on a 4 point scale that consisted of score from 0-3 where, 0=would never dose, 1=slight chance of dozing, 2=moderate chance of dozing, 3=high chance of dozing). The total ESS score is sum of scores on 8 items. Last assessed value of OLP (Day 28) value was used as baseline value for DBP. Change from end of OLP was calculated by subtracting the value on Day 28 minus the value on Day 42.
Change from Baseline in the Leeds Sleep Evaluation Questionnaire (LSEQ) during the OLP | Baseline (Day -1) up to Day 28
  The LSEQ had 10 questions captured on a 100mm VAS which allowed qualitative assessment of sleep. Four domain scores were calculated: 1. Getting to Sleep (GTS)-1. Easier than usual/Harder than usual, 2. Quicker than usual/Slower than usual or 3. Felt more drowsy than usual/Felt less drowsy than usual (Average of 1, 2, 3); 2. Quality of Sleep (QOS)- 4. More restful than usual/More restless than usual or 5. Fewer periods of wakefulness than usual/More periods of wakefulness than usual (Average 4 and 5); 3. Awakening from Sleep (AFS)- 6. Easier than usual/More difficult than usual or 7. Took shorter than usual/Took longer than usual (Average of 6 and 7); 4. Behavior Following Waking (BFW)- 8 and 9. Alert/Tired or 10. Less clumsy than usual/More clumsy than usual (Average of 8, 9 and 10). Baseline was defined at Visit 1 (Day -1). Change from baseline was calculated by subtracting the value on Day -1 minus the value on Day 1-6,7-13,14-20,21-29.
Change from End of OLP in the LSEQ during the DBP | Day 28 up to Day 42
  The LSEQ had 10 questions captured on a 100mm VAS which allowed qualitative assessment of sleep. Four domain scores were calculated: 1. Getting to Sleep (GTS)-1. Easier than usual/Harder than usual, 2. Quicker than usual/Slower than usual or 3. Felt more drowsy than usual/Felt less drowsy than usual (Average of 1, 2, 3); 2. Quality of Sleep (QOS)- 4. More restful than usual/More restless than usual or 5. Fewer periods of wakefulness than usual/More periods of wakefulness than usual (Average 4 and 5); 3. Awakening from Sleep (AFS)- 6. Easier than usual/More difficult than usual or 7. Took shorter than usual/Took longer than usual (Average of 6 and 7); 4. Behavior Following Waking (BFW)- 8 and 9. Alert/Tired or 10. Less clumsy than usual/More clumsy than usual (Average of 8, 9, and 10). Last assessed value of OLP (Day 28) value was used as baseline value for DBP. Change from end of OLP was calculated by subtracting the value on Day 28 minus the value on Day 30-35 and Day 36-42.
Change from Baseline in Frequency of Daytime Naps (Based on Actigraphy) during the OLP | Baseline up to Day 28
  The number of daytime naps was calculated based on Actigraphy. Actigraphy data was collected using the Actiwatch activity monitoring system. Participants were asked to continuously wear a small actigraphy monitor on the wrist of their non-dominant arm during the study in order to objectively monitor sleep quality and daytime napping. The Actiwatch was a wrist-worn device that produced a signal as the wearer made physical movement which was used as a surrogate marker of sleep. Participants marked time in bed manually with the watch, which improved assessment of sleep efficiency. Baseline was defined at Visit 1 (Day -7). Change from baseline was calculated by subtracting the value on Day -7 minus the value on Day 1-6,7-13,14-20,21-29.
Change from Baseline in duration of Daytime Naps (Based on Actigraphy) during the OLP | Baseline up to Day 28
  The duration of daytime naps was calculated based on Actigraphy. Actigraphy data was collected using the Actiwatch activity monitoring system. Participants were asked to continuously wear a small actigraphy monitor on the wrist of their non-dominant arm during the study in order to objectively monitor sleep quality and daytime napping. The Actiwatch was a wrist-worn device that produced a signal as the wearer made physical movement which was used as a surrogate marker of sleep. Participants marked time in bed manually with the watch, which improved assessment of sleep efficiency. Baseline was defined at Visit 1 (Day -7). Change from baseline was calculated by subtracting the value on Day -7 minus the value on Day 1-6,7-13,14-20,21-29.
Change from End of OLP (Day 28) in Frequency of Daytime Naps (Based on Actigraphy) during the DBP | Day 28 up to Day 42
  The number of daytime naps was calculated based on Actigraphy. Actigraphy data was collected using the Actiwatch activity monitoring system. Participants were asked to continuously wear a small actigraphy monitor on the wrist of their non-dominant arm during the study in order to objectively monitor sleep quality and daytime napping. The Actiwatch was a wrist-worn device that produced a signal as the wearer made physical movement which was used as a surrogate marker of sleep. Participants marked time in bed manually with the watch, which improved assessment of sleep efficiency. Last assessed value of OLP (Day 28) value was used as baseline value for DBP. Change from end of OLP was calculated by subtracting the value on Day 28 minus the value on Day 30-35 and Day 36-42. Least square mean was used to present the value for adjusted mean.
Change from End of OLP (Day 28) in duration of Daytime Naps (Based on Actigraphy) during the DBP | Day 28 up to Day 42
  The duration of daytime naps was calculated based on Actigraphy. Actigraphy data was collected using the Actiwatch activity monitoring system. Participants were asked to continuously wear a small actigraphy monitor on the wrist of their non-dominant arm during the study in order to objectively monitor sleep quality and daytime napping. The Actiwatch was a wrist-worn device that produced a signal as the wearer made physical movement which was used as a surrogate marker of sleep. Participants marked time in bed manually with the watch, which improved assessment of sleep efficiency. Last assessed value of OLP (Day 28) value was used as baseline value for DBP. Change from end of OLP was calculated by subtracting the value on Day 28 minus the value on Day 30-35 and Day 36-42. Least square mean was used to present the value for adjusted mean.
Number of participants who responded to open-label treatment on Day 28 | Day 28
  The number of participants who responded to treatment at the end of the OLP (Day 28) and who were randomized to the DBP have been presented. Treatment response was defined as a 2 minute increase in sleep latency in the MWT from baseline and a sleep latency in the MWT of at least 5 minutes on Day 28.
Change from Baseline in Time (min) until Sleep Onset REM (rapid eye moment) (SOREM) during the OLP | Baseline (Day -1) up to Day 28
  In normal participants, the sleep cycle comprised of 3 to 4 stages of slow-wave or non-REM (NREM) sleep lasting about 90 min. Each NREM sleep period was followed by a period of REM sleep i.e. it was necessary to pass through the non-REM cycle to enter into the REM state. REM sleep was characterized by increased brain activity, dreaming and loss of muscle tone i.e. REM sleep atonia. In narcolepsy, the cycle of NREM alternating with REM was abnormal and entry occured directly into REM sleep with a latency to onset of REM sleep that was abnormally shortened (sleep onset REM). REM sleep was characterised by increased brain activity, dreaming and loss of muscle tone i.e. REM sleep atonia. SOREM was measured on overnight Polysomnography (PSG) used to assess sleep architecture. Baseline was defined at Day -1. Change from baseline was calculated by subtracting the value on Day -1 minus the value on Day 13 and 27.
Change from End of OLP in Time (min) until SOREM to the End of DBP | Day 28 and Day 42
  In normal participants, sleep cycle comprised of 3 to 4 stages of slow-wave or non-REM (NREM) sleep lasting about 90 min. Each NREM sleep period was followed by period of REM sleep i.e. it was necessary to pass through non-REM cycle to enter into REM state. REM sleep was characterized by increased brain activity,dreaming and loss of muscle tone i.e. REM sleep atonia. In narcolepsy, cycle of NREM alternating with REM was abnormal and entry occured directly into REM sleep with a latency to onset of REM sleep that was abnormally shortened (sleep onset REM). REM sleep was characterised by increased brain activity, dreaming and loss of muscle tone i.e. REM sleep atonia. SOREM was measured on overnight PSG which was used to assess sleep architecture. Last assessed value of OLP (Day 28) value was used as baseline value for DBP. Change from end of OLP was calculated by subtracting the value on Day 28 minus the value on Day 42. Least square mean was used to present the value for adjusted mean.
Number of participants with Improved assessment of illness on day 14 and 28 as measured by the Patient Global Impression of Change (PGIC) and by the Clinician Global Impression of Change (CGIC) | Day 14 and 28
  Disease severity was scored by the clinician (CGIC) and participant (PGIC) using a verbal rating scale from 1-7 which was as follows: 1.Very much improved, 2.Much improved, 3.Minimally improved, 4.No change, 5.Minimally worse, 6.Much worse and 7.Very much worse. During OLP (until Day 28), the investigator/participant indicated their assessment of total improvement or worsening compared with the same participant's condition at start of treatment, whether or not the change was due to drug. However, when disease severity was assessed at end of DBP, the assessor rated any change in disease severity recorded at the beginning of DBP (Day 28), rather than the start of treatment. At this time, participants randomised to active treatment were expected to have "No change" or perhaps a minimal change, while participants randomised to placebo were expected to have answers such as "Much worse" or "Very much worse", demonstrating a loss of response upon active treatment withdrawal.
Number of participants with Improved assessment of illness on day 42 as measured by the PGIC and by the CGIC | Day 42
  Disease severity was scored by the clinician (CGIC) and participant (PGIC) using a verbal rating scale from 1-7 which was as follows: 1.Very much improved, 2.Much improved, 3.Minimally improved, 4.No change, 5.Minimally worse, 6.Much worse and 7.Very much worse. During OLP (until Day 28), the investigator/participant indicated their assessment of total improvement or worsening compared with the same participant's condition at start of treatment, whether or not the change was due to drug. However, when disease severity was assessed at end of DBP, the assessor rated any change in disease severity recorded at the beginning of DBP (Day 28), rather than the start of treatment. At this time, participants randomised to active treatment were expected to have "No change" or perhaps a minimal change, while participants randomised to placebo were expected to have answers such as "Much worse" or "Very much worse", demonstrating a loss of response upon active treatment withdrawal.
Change from Baseline in Time (min) required to complete the Digit Vigilance Test (DVT) during the OLP | Baseline (Day -1) up to Day 28
  Participants completed the two-page DVT at the end of each MWT assessment. Participants were required to scan through two pages of numbers and cross out every time the control number (either a 6 or a 9) appeared. The total time taken to complete the task was recorded. Baseline was defined at Visit 1 (Day -1). Change from baseline was calculated by subtracting the value on Day -1 minus the value on Day 14 and 28.
Change from End of OLP in Time (min) Required to Complete the DVT during the DBP (Day 42) | Day 28 and Day 42
  Participants completed the two-page DVT at the end of each MWT assessment. Participants were required to scan through two pages of numbers and cross out every time the control number (either a 6 or a 9) appeared. The total time taken to complete the task was recorded. Last assessed value of OLP (Day 28) value was used as baseline value for DBP. Change from end of OLP was calculated by subtracting the value on Day 28 minus the value on Day 42. Least square mean was used to present the value for adjusted mean.
Change from Baseline in number of errors on the DVT to the End of OLP (Day 28) | Baseline (Day -1), Day 14 and Day 28
  Participants completed the two-page DVT at the end of each MWT assessment. Participants were required to scan through two pages of numbers and cross out every time the control number (either a 6 or a 9) appeared. The percent accuracy (number of errors) to complete the task was recorded. Baseline was defined at Visit 1 (Day -1). Change from baseline was calculated by subtracting the value on Day -1 minus the value on Day 14 and 28.
Change from End of OLP (Day 28) in number of errors on the DVT to the End of DBP (Day 42) | Day 28 and Day 42
  Participants completed the two-page DVT at the end of each MWT assessment. Participants were required to scan through two pages of numbers and cross out every time the control number (either a 6 or a 9) appeared. The percent accuracy (number of errors) to complete the task was recorded. Last assessed value of OLP (Day 28) value was used as baseline value for DBP. Change from end of OLP was calculated by subtracting the value on Day 28 minus the value on Day 42. Least square mean was used to present the value for adjusted mean.
Change from baseline in Vital Signs for the OLP- Systolic blood pressure and diastolic blood pressure | Baseline (Day 1) up to Day 28
  Safety assessment was performed for systolic and diastolic blood pressure on Day 1 (4,8,12 hour post-dose), 7 (4,8,12 hour post-dose), 14 (4,8,12 hour post-dose), 21 (4,8,12 hour post-dose) and 28 (prior to sleep test 1,2,3,4) during the OLP. Blood pressure (systolic and diastolic) was recorded in semi-supine position. Measurements were made after the participant had been resting semi-supine for a period of at least 3 minutes. During the resting period the participants were supervised to ensure they did not fall asleep. Baseline was defined as the mean of the 3 pre-dose assessments taken on Day 1. Change from Baseline was calculated by subtracting the value on Day 1 minus the value on Day 1, 7, 14, 21 and 28.
Change from baseline in Vital Signs for the DBP- Systolic blood pressure and diastolic blood pressure | Baseline (Day 1) and Day 42
  Safety assessment was performed for systolic and diastolic blood pressure on Day 42 (prior to sleep test 1, 2, 3 and 4) during the DBP. Blood pressure (systolic and diastolic) was recorded in semi-supine position. Measurements were made after the participant had been resting semi-supine for a period of at least 3 minutes. During the resting period the participants were supervised to ensure they did not fall asleep. Baseline was defined as the mean of the 3 pre-dose assessments taken on Day 1. Change from Baseline was calculated by subtracting the value on Day 1 minus the value on Day 42.
Change from baseline in Vital Signs for the OLP- Heart rate (HR) | Baseline (Day 1) up to Day 28
  Safety assessment was performed for HR on Day 1 (pre dose, 4, 8 and 12 hour post dose), 7 (pre dose, 4, 8 and 12 hour post dose), 14 (pre dose, 4, 8 and 12 hour post dose), 21 (pre dose, 4, 8 and 12 hour post dose) and 28 (prior to sleep test 1, 2, 3 and 4) during the OLP. Heart rate was recorded in semi-supine position. Measurements were made after the participant had been resting semi-supine for a period of at least 3 minutes. During the resting period the participants were supervised to ensure they did not fall asleep. Baseline was defined as the mean of the 3 pre-dose assessments taken on Day 1. Change from Baseline was calculated by subtracting the value on Day 1 minus the value on Day 1, 7, 14, 21 and 28.
Change from baseline in Vital Signs for the DBP- HR | Baseline (Day 1) and Day 42
  Safety assessment was performed for HR on Day 42 (prior to sleep test 1, 2, 3 and 4) during the DBP. Heart rate was recorded in semi-supine position. Measurements were made after the participant had been resting semi-supine for a period of at least 3 minutes. During the resting period the participants were supervised to ensure they did not fall asleep. Baseline was defined as the mean of the 3 pre-dose assessments taken on Day 1. Change from Baseline was calculated by subtracting the value on Day 1 minus the value on Day 42.
Number of participants with abnormal electrocardiogram (ECG) findings at any time during OLP | Up to Day 28
  All ECGs were recorded after at least 3 minutes rest in a semi-supine position. During this resting period, participants were supervised to ensure they did not fall asleep. Where possible, hot or cold drinks and food was avoided 30 minutes before an ECG measurement. All ECGs were recorded after at least 3 minutes rest in a semi-supine position. Data for any OLP post baseline was reported for abnormal-not clinically significant (NCS) values.
Number of participants with abnormal ECG findings during DBP | Day 42
  All ECGs were recorded after at least 3 minutes rest in a semi-supine position. During this resting period, participants were supervised to ensure they did not fall asleep. Where possible, hot or cold drinks and food was avoided 30 minutes before an ECG measurement. All ECGs were recorded after at least 3 minutes rest in a semi-supine position. Data for Day 42 prior to sleep test 1, 2, 3 and 4 was reported for abnormal- NCS.
Change from Baseline in Profile of Mood State (POMS-B) Domain Scores for the OLP | Baseline (Day -1) up to Day 28
  POMS scale was an adjective rating scale and considered to be a standardized mood-state inventory. The short form of the POMS was a 30 word-item questionnaire that was completed by the participant. Participants were instructed to rate each adjective on the basis of how they felt at the present time on a scale. The short form consisted of 30 adjective words with 5-point scale degrees of agreement (0=applies not at all, 4=applies extremely) and yielded six types of mood states: tension-anxiety (sum of 1, 6, 12, 16, and 20), depression-dejection (sum of 7, 11, 15, 17, and 21), anger-hostility (sum of 2, 9, 14, 25, and 28), vigour-activity (sum of 4, 8, 10, 27, and 30), fatigue-inertia (sum of 3, 13, 19, 22, and 23) and confusion-bewilderment (sum of 5, 18, 24, 26, and 29). Baseline was defined at Visit 1 (Day -1). Change from baseline was calculated by subtracting the value on Day -1 minus the value on Day 14 and 28.
Change from Baseline in POMS-B Domain Scores for the DBP | Baseline (Day -1) up to Day 42
  POMS scale was an adjective rating scale and considered to be a standardized mood-state inventory. The short form of the POMS was a 30 word-item questionnaire that was completed by the participant. Participants were instructed to rate each adjective on the basis of how they felt at the present time on a scale. The short form consisted of 30 adjective words with 5-point scale degrees of agreement (0=applies not at all, 4=applies extremely) and yielded six types of mood states: tension-anxiety (sum of 1, 6, 12, 16, and 20), depression-dejection (sum of 7, 11, 15, 17, and 21), anger-hostility (sum of 2, 9, 14, 25, and 28), vigour-activity (sum of 4, 8, 10, 27, and 30), fatigue-inertia (sum of 3, 13, 19, 22, and 23) and confusion-bewilderment (sum of 5, 18, 24, 26, and 29). Baseline was defined at Visit 1 (Day -1). Change from Baseline was calculated by subtracting the value on Day -1 minus the value on Day 42.
Assessment of Nocturnal Actigraphy for the OLP- Average actual sleep time, Average actual wake time, Average sleep latency duration | Day 28
  Actigraphy data was collected using the Actiwatch activity monitoring system. Participants were asked to continuously wear a small actigraphy monitor on the wrist of their non-dominant arm during the study in order to objectively monitor sleep quality and daytime napping. The Actiwatch was a wrist-worn device that produced a signal as the wearer makes physical movement which was used as a surrogate marker of sleep. Participants marked time in bed manually with the watch, which improved assessment of sleep efficiency. Nocturnal actigraphy parameters summarized for this outcome measure was average actual sleep time, average actual wake time and average sleep latency duration. Actigraphy was performed on Day -7 to -1, 1 to 6, 7 to 13, 14 to 20 and 21 to 29 during the OLP.
Assessment of Nocturnal Actigraphy for the OLP- Average sleep efficiency | Up to Day 28
  Actigraphy data was collected using the Actiwatch activity monitoring system. Participants were asked to continuously wear a small actigraphy monitor on the wrist of their non-dominant arm during the study in order to objectively monitor sleep quality and daytime napping. The Actiwatch was a wrist-worn device that produced a signal as the wearer makes physical movement which was used as a surrogate marker of sleep. Participants marked time in bed manually with the watch, which improved assessment of sleep efficiency. Nocturnal actigraphy parameter summarized for this outcome measure was average sleep efficiency. Actigraphy was performed on Day -7 to -1, 1 to 6, 7 to 13, 14 to 20 and 21 to 29 during the OLP.
Assessment of Nocturnal Actigraphy for the DLP- Average actual sleep time, Average actual wake time, Average sleep latency duration | Up to Day 42
  Actigraphy data was collected using the Actiwatch activity monitoring system. Participants were asked to continuously wear a small actigraphy monitor on the wrist of their non-dominant arm during the study in order to objectively monitor sleep quality and daytime napping. The Actiwatch was a wrist-worn device that produced a signal as the wearer makes physical movement which was used as a surrogate marker of sleep. Participants marked time in bed manually with the watch, which improved assessment of sleep efficiency. Nocturnal actigraphy parameters summarized for this outcome measure was average actual sleep time, average actual wake time and average sleep latency duration. Actigraphy was performed on Day 30 to 35 and 36 to 42 during the DBP.
Assessment of Nocturnal Actigraphy for the DLP- Average sleep efficiency | Up to Day 42
  Actigraphy data was collected using the Actiwatch activity monitoring system. Participants were asked to continuously wear a small actigraphy monitor on the wrist of their non-dominant arm during the study in order to objectively monitor sleep quality and daytime napping. The Actiwatch was a wrist-worn device that produced a signal as the wearer makes physical movement which was used as a surrogate marker of sleep. Participants marked time in bed manually with the watch, which improved assessment of sleep efficiency. Nocturnal actigraphy parameters summarized for this outcome measure was a average sleep efficiency. Actigraphy was performed on Day 30 to 35 and 36 to 42 during the DBP.
Change from Baseline in Nocturnal PSG for the OLP- Frequency of awakening | Baseline (Day -1) up to Day 28
  PSG was used to assess sleep architecture. Nocturnal PSG was recorded as a safety measure at Baseline (Day -1), Day 13 and Day 27. Variables that describe sleep architecture include total sleep time, sleep efficiency, sleep latency, latencies to each sleep stage, time spent in each sleep stage, etc. The PSG parameter summarized for this outcome measure was frequency of awakening (count). Baseline was defined at Visit 1 (Day -1). Change from Baseline was calculated by subtracting the value on Day -1 minus the value on Day 13 and 27.
Change from Baseline in Nocturnal PSG for the OLP- total movement time, REM duration (REM-D), REM-D in first, second, third and fourth quarter of sleep, REM latency | Baseline (Day -1) up to Day 28
  PSG was used to assess sleep architecture. Nocturnal PSG was recorded as a safety measure at Baseline (Day -1), Day 13 and Day 27. Variables that describe sleep architecture include total sleep time, sleep efficiency, sleep latency, latencies to each sleep stage, time spent in each sleep stage, etc. The PSG parameter summarized for this outcome measure were total movement time, REM-D, REM-D in first, second, third and fourth quarter of sleep and REM latency. Baseline was defined at Visit 1 (Day -1). Change from Baseline was calculated by subtracting the value on Day -1 minus the value on Day 13 and 27.
Change from Baseline in Nocturnal PSG for the OLP- Sleep efficiency | Baseline (Day -1) up to Day 28
  PSG was used to assess sleep architecture. Nocturnal PSG was recorded as a safety measure at Baseline (Day -1), Day 13 and Day 27. Variables that describe sleep architecture include total sleep time, sleep efficiency, sleep latency, latencies to each sleep stage, time spent in each sleep stage, etc. The PSG parameter summarized for this outcome measure was sleep efficiency. Baseline was defined at Visit 1 (Day -1). Change from Baseline was calculated by subtracting the value on Day -1 minus the value on Day 13 and 27.
Change from Baseline in Nocturnal PSG for the OLP- Sleep onset latency, Sleep period time, total Stage 1, 2, 3, 4 duration | Baseline (Day -1) up to Day 28
  PSG was used to assess sleep architecture. Nocturnal PSG was recorded as a safety measure at Baseline (Day -1), Day 13 and Day 27. Variables that describe sleep architecture include total sleep time, sleep efficiency, sleep latency, latencies to each sleep stage, time spent in each sleep stage, etc. The PSG parameter summarized for this outcome measure was Sleep onset latency, Sleep period time, total Stage 1, 2, 3, 4 duration. Baseline was defined at Visit 1 (Day -1). Change from Baseline was calculated by subtracting the value on Day -1 minus the value on Day 13 and 27.
Change from Baseline in Nocturnal PSG for the OLP- Time in bed, Total sleep time, Wake during sleep (WDS) from first epoch of sleep (SO) to final epoch of sleep | Baseline (Day -1) up to Day 28
  PSG was used to assess sleep architecture. Nocturnal PSG was recorded as a safety measure at Baseline (Day -1), Day 13 and Day 27. Variables that describe sleep architecture include total sleep time, sleep efficiency, sleep latency, latencies to each sleep stage, time spent in each sleep stage, etc. The PSG parameter summarized for this outcome measure was Time in bed, Total sleep time and WDS from SO to final epoch of sleep. Baseline was defined at Visit 1 (Day -1). Change from Baseline was calculated by subtracting the value on Day -1 minus the value on Day 13 and 27.
Change from Baseline in Nocturnal PSG for the DBP- Frequency of awakening | Baseline (Day -1) and Day 42
  PSG was used to assess sleep architecture. Nocturnal PSG was recorded as a safety measure at Baseline (Day -1) and Day 42. Variables that describe sleep architecture include total sleep time, sleep efficiency, sleep latency, latencies to each sleep stage, time spent in each sleep stage, etc. The PSG parameter summarized for this outcome measure was frequency of awakening (count). Baseline was defined at Visit 1 (Day -1). Change from Baseline was calculated by subtracting the value on Day -1 minus the value on Day 42.
Change from Baseline in Nocturnal PSG for the DBP- total movement time, REM-D, REM-D in first, second, third and fourth quarter of sleep, REM latency | Baseline (Day -1) and Day 42
  PSG was used to assess sleep architecture. Nocturnal PSG was recorded as a safety measure at Baseline (Day -1) and Day 42. Variables that describe sleep architecture include total sleep time, sleep efficiency, sleep latency, latencies to each sleep stage, time spent in each sleep stage, etc. The PSG parameter summarized for this outcome measure was total movement time, REM-D, REM-D in first, second, third and fourth quarter of sleep and REM latency. Baseline was defined at Visit 1 (Day -1). Change from Baseline was calculated by subtracting the value on Day -1 minus the value on Day 42.
Change from Baseline in Nocturnal PSG for the DBP- Sleep efficiency | Baseline (Day -1) and Day 42
  PSG was used to assess sleep architecture. Nocturnal PSG was recorded as a safety measure at Baseline (Day -1), Day 42. Variables that describe sleep architecture include total sleep time, sleep efficiency, sleep latency, latencies to each sleep stage, time spent in each sleep stage, etc. The PSG parameter summarized for this outcome measure was sleep efficiency. Baseline was defined at Visit 1 (Day -1). Change from Baseline was calculated by subtracting the value on Day -1 minus the value on Day 42.
Change from Baseline in Nocturnal PSG for the DBP- Sleep onset latency, Sleep period time, total Stage 1, 2, 3, 4 duration | Baseline (Day -1) and Day 42
  PSG was used to assess sleep architecture. Nocturnal PSG was recorded as a safety measure at Baseline (Day -1) Day 42. Variables that describe sleep architecture include total sleep time, sleep efficiency, sleep latency, latencies to each sleep stage, time spent in each sleep stage, etc. The PSG parameter summarized for this outcome measure was Sleep onset latency, Sleep period time, total Stage 1, 2, 3, 4 duration. Baseline was defined at Visit 1 (Day -1). Change from Baseline was calculated by subtracting the value on Day -1 minus the value on Day 42.
Change from Baseline in Nocturnal PSG for the DBP- Time in bed, Total sleep time, WDS from SO to final epoch of sleep | Baseline (Day -1) and Day 42
  PSG was used to assess sleep architecture. Nocturnal PSG was recorded as a safety measure at Baseline (Day -1) Day 42. Variables that describe sleep architecture include total sleep time, sleep efficiency, sleep latency, latencies to each sleep stage, time spent in each sleep stage, etc. The PSG parameter summarized for this outcome measure was Time in bed, Total sleep time and WDS from SO to final epoch of sleep. Baseline was defined at Visit 1 (Day -1). Change from Baseline was calculated by subtracting the value on Day -1 minus the value on Day 42.
Number of participants with shift from Baseline in haematology parameters of potential clinical importance (PCI) for OLP | Baseline (Day 1) up to Day 28
  Blood samples were taken for analysis of white blood cell count (WBC) (normal range [NR]: 3.8-10.8 giga cells/liter [GI/L]), red blood cell count (RBC) (NR: 4.4-5.8 trillion cells/liter [TI/L]), haemoglobin (Hb) (NR: 138-172 gram/liter [G/L]), haematocrit (HCT) (NR: 0.41-0.5 L), mean cell volume (MCV) (NR: 80-100 femto liter [FL]), mean cell haemoglobin (MCH) (NR: 27-33 picograms [PG]), mean cell haemoglobin concentration (MCHC) (NR: 320-360 G/L), platelet count (130-400 GI/L), segmented neutrophil count (SN) (NR: 1.8-8 GI/L), lymphocyte count (NR: 0.85-4.1 GI/L), monocyte count (NR: 0.2-1.1 GI/L), eosinophil count (NR: 0.05-0.55 GI/L) and basophil count (NR: 0-0.2 GI/L). Data for participants with a shift in values from Baseline (PCI high, within range (WR) and PCI low) to Day 7, 14, 21 and 28 was reported. Baseline (defined at Day 1 pre-dose) was the mean of the 3 pre-dose assessments taken on Day 1.
Number of participants with shift from baseline in Haematology parameters of PCI for DBP | Baseline (Day 1) up to Day 42
  Blood samples were taken for analysis of WBC (NR: 3.8-10.8 GI/L), RBC (NR: 4.4-5.8 TI/L), Hb (NR: 138-172 G/L), HCT (NR: 0.41-0.5 L), MCV (NR: 80-100 FL), MCH (NR: 27-33 PG), MCHC (NR: 320-360 G/L), platelet count (130-400 GI/L), SN (NR: 1.8-8 GI/L), lymphocyte count (NR: 0.85-4.1 GI/L), monocyte count (NR: 0.2-1.1 GI/L), eosinophil count (NR: 0.05-0.55 GI/L) and basophil count (NR: 0-0.2 GI/L). Data for participants with a shift in values from Baseline (PCI high, WR and PCI low) to Day 42 was reported. Baseline (defined at Day 1 pre-dose) was the mean of the 3 pre-dose assessments taken on Day 1.
Number of participants with shift from baseline in clinical chemistry parameters of PCI for OLP | Baseline (Day 1) up to day 28
  Blood samples were taken for the analysis of Alkaline phosphatase (20 - 125 international units/liter [IU/L]), Alanine transaminase (ALT) (0 - 48 IU/L), Aspartate transaminase (AST) (0 - 42 IU/L), Gamma-glutamyl transpeptidase (GGT) (0 - 65 IU/L), Glucose (3.9 - 6.9 mmol/L), Cholesterol (0 - 5.15 mmol/L), Triglycerides (0 - 2.24 mmol/L), Albumin (32 - 50 G/L), Total protein (60 - 85 G/L), Total bilirubin (0 - 22 UMOL/L), Creatinine (44 - 124 UMOL/L), Creatine phosphokinase (0 - 235 IU/L), Sodium (135 - 146 MMOL/L), Potassium (3.5 - 5.3 MMOL/L), Chloride (95 - 108 MMOL/L), Calcium (2.12 - 2.56 MMOL/L), Urea (2.5 - 9 MMOL/L), TSH, Thyroxine (T3) (10.3 - 23.2 PMOL/L) and T4. The number of participants with values outside pre-determined clinically important ranges, i.e., values of PCI was reported for Day 7, 14, 21, 28. Baseline (defined at Day 1 pre-dose) was the mean of the 3 pre-dose assessments taken on Day 1.
Number of participants with shift from Baseline in clinical chemistry parameters of PCI for DBP | Baseline (Day 1) up to Day 42
  Blood samples were taken for the analysis of Alkaline phosphatase (20 - 125 international units/liter [IU/L]), Alanine transaminase (ALT) (0 - 48 IU/L), Aspartate transaminase (AST) (0 - 42 IU/L), Gamma-glutamyl transpeptidase (GGT) (0 - 65 IU/L), Glucose (3.9 - 6.9 mmol/L), Cholesterol (0 - 5.15 mmol/L), Triglycerides (0 - 2.24 mmol/L), Albumin (32 - 50 G/L), Total protein (60 - 85 G/L), Total bilirubin (TL) (0 - 22 UMOL/L), Creatinine (44 - 124 UMOL/L), Creatine phosphokinase (0 - 235 IU/L), Sodium (135 - 146 MMOL/L), Potassium (3.5 - 5.3 MMOL/L), Chloride (95 - 108 MMOL/L), Calcium (2.12 - 2.56 MMOL/L), Urea (2.5 - 9 MMOL/L), TSH, Thyroxine (T3) (10.3 - 23.2 PMOL/L) and T4. The number of participants with values outside pre-determined clinically important ranges, i.e., values of PCI was reported for Day 42. Baseline (defined at Day 1 pre-dose) was the mean of the 3 pre-dose assessments taken on Day 1.
Number of participants with adverse events (AEs) and serious adverse events (SAEs) in the OLP | Up to Day 28
  AE was defined as any untoward medical occurrence in a participant , temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE was any untoward medical occurrence that, at any dose: results in death, was life threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect or was considered as medically significant. No SAEs were reported in this study.
Number of participants with AEs and SAEs in the DBP | Up to Day 42
  AE was defined as any untoward medical occurrence in a participant , temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE was any untoward medical occurrence that, at any dose: results in death, was life threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect or was considered as medically significant. No SAEs were reported in this study.
Number of participants with abnormal urinalysis results for the OLP | Up to Day 28
  Approximately 10-20 milliliter (mL) mid-stream urine was collected into a sterile container and it was tested for protein, glucose, ketones, bilirubin, blood, urobilinogen and leucocytes during Baseline, Day 7, 14, 21 and 28. Sediment microscopy was performed only when any of the tests were abnormal, in such cases microscopy was performed for WBC (Urine Leukocyte Esterase test [ULET] for detecting WBC), RBC, Hyaline casts, Granular casts and Cellular casts. Urinalysis result was considered 'positive' when there was any amount of blood or protein, etc. detected in the urine sample. Any blood or protein that was detected was referred to as an 'abnormality'.
Number of participants with abnormal urinalysis results for the DBP | Day 42
  Approximately 10-20 mL mid-stream urine was collected into a sterile container and it was tested for protein, glucose, ketones, bilirubin, blood, urobilinogen and leucocytes during DBP (Day 42). Sediment microscopy was performed only when any of the tests were abnormal, in such cases microscopy was performed for WBC (ULET for detecting WBC), RBC, Hyaline casts, Granular casts and Cellular casts. Urinalysis result was considered 'positive' when there was any amount of blood or protein, etc. detected in the urine sample. Any blood or protein that was detected was referred to as an 'abnormality'.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- Austria (2):
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Vienna
- GSK Investigational Site, Espoo, Finland
- Germany (5):
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Schwalmstadt, Hesse
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Berlin, State of Berlin
- GSK Investigational Site, Leiden, Netherlands
- GSK Investigational Site, Barcelona, Spain
- United Kingdom (3):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, London, London
  - GSK Investigational Site, Edinburgh